CLINICAL TRIAL: NCT00989287
Title: Safety and Immunogenicity Study of GSK Biologicals' Influenza Vaccine GSK2340272A in Adults Aged 18 to 60 Years
Brief Title: Immunogenicity and Safety Study of an Investigational Influenza (H1N1 Influenza Virus) Vaccine in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 113866; 2009-016078-33 (EudraCT Number)
Record Dates: First submitted 2009-10-01; First posted 2009-10-05 (Estimated); Results first posted 2018-03-05 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Influenza
Keywords: GSK Bio's influenza vaccine GSK2340272A; influenza infection
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- GSK2340272A Group (Experimental): Healthy male or female adults, between and including 18 to 60 years of age, who received two doses of GSK2340272A vaccine, administered intramuscularly in the deltoid region of the non-dominant arm at Day 0 and of the dominant arm at Day 21.
  Interventions: Biological: GSK2340272A
- GSK2340269A Group (Experimental): Healthy male or female adults, between and including 18 to 60 years of age, who received two doses of GSK2340269A vaccine, administered intramuscularly in the deltoid region of the non-dominant arm at Day 0 and of the dominant arm at Day 21.
  Interventions: Biological: GSK2340269A

INTERVENTIONS:
Biological: GSK2340272A — Two intramuscular injections in the deltoid region of the non-dominant arm.
  Arms: GSK2340272A Group
Biological: GSK2340269A — Two intramuscular injections in the deltoid region of the non-dominant arm.
  Arms: GSK2340269A Group

SUMMARY:
The objective of this study is to evaluate the immunogenicity and safety of GSK Biologicals' investigational vaccine GSK2340272A in adults aged 18 to 60 years.

DETAILED DESCRIPTION:
This Protocol Posting has been updated following Protocol amendment 1, October 2009. The impacted section is the outcomes measures section.

ELIGIBILITY:
Inclusion Criteria:

* A male or female aged 18 to 60 years at the time of the first vaccination.
* Subjects who the investigator believes that they can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject.
* Satisfactory baseline medical assessment by history and physical examination. Stable health status is defined as the absence of health event satisfying the definition of an SAE, or a change in an ongoing drug therapy due to therapeutic failure or symptoms of drug toxicity, within one month prior to enrolment.
* Access to a consistent means of telephone contact, which may be either in the home or at the workplace, land line or mobile, but NOT a pay phone or multiple-user device.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject: has practiced adequate contraception for 30 days prior to vaccination, and has a negative pregnancy test on the day of vaccination, and has agreed to continue adequate contraception during the entire treatment period and for two months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of the study vaccine or planned use during the study period. Potential subjects in the follow-up phase of a prior investigational study may be enrolled if the investigator's judgment is that it will have no effect on safety, reactogenicity, or immunogenicity endpoints in this study, and that it does not violate the protocol requirements of the prior trial.
* Presence of evidence of substance abuse or of neurological or psychiatric diagnoses which, although stable, are deemed by the investigator to render the potential subject unable/unlikely to provide accurate safety reports.
* Presence of an axillary temperature >= 37.5°C, or acute symptoms greater than "mild" severity on the scheduled date of first vaccination.
* Diagnosed with cancer, or treatment for cancer, within the past three years.
* Any confirmed or suspected immunosuppressive or immunodeficient condition including history of human immunodeficiency virus (HIV) infection.
* Clinically or virologically confirmed influenza infection within six months preceding the study start.
* Chronic administration of immunosuppressants or other immune modifying drugs within six months of study enrolment or planned administration during the study period. For corticosteroids, this will mean a dose equivalent to 20 mg/day of prednisone or equivalent for persons for > two weeks. Inhaled and topical steroids are allowed.
* Receipt of any immunoglobulins and/or any blood products within three months of study enrolment or planned administration of any of these products during the study period.
* Any significant disorder of coagulation or treatment with warfarin derivatives or heparin. Persons receiving individual doses of low molecular weight heparin outside of 24 hours prior to vaccination are eligible. Persons receiving prophylactic antiplatelet medications and without a clinically-apparent bleeding tendency, are eligible.
* An acute evolving neurological disorder or history of Guillain-Barré syndrome.
* Administration of any vaccines within 30 days before vaccination.
* Any known or suspected allergy to any constituent of influenza vaccines; a history of anaphylactic-type reaction to any constituent of influenza vaccines; or a history of severe adverse reaction to a previous influenza vaccine.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* Any conditions which, in the opinion of the investigator, prevents the subjects from participating in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 131 (Actual)
Dates: Start 2009-10-07 (Actual); Primary Completion 2009-10-09 (Actual); Study Completion 2010-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Background] Roman F, Clement F, Dewe W, Walravens K, Maes C, Willekens J, De Boever F, Hanon E, Leroux-Roels G. Effect on cellular and humoral immune responses of the AS03 adjuvant system in an A/H1N1/2009 influenza virus vaccine administered to adults during two randomized controlled trials. Clin Vaccine Immunol. 2011 May;18(5):835-43. doi: 10.1128/CVI.00480-10. Epub 2011 Mar 30. PMID 21450978
- [Derived] van der Most RG, Clement F, Willekens J, Dewe W, Walravens K, Vaughn DW, Leroux-Roels G. Long-Term Persistence of Cell-Mediated and Humoral Responses to A(H1N1)pdm09 Influenza Virus Vaccines and the Role of the AS03 Adjuvant System in Adults during Two Randomized Controlled Trials. Clin Vaccine Immunol. 2017 Jun 5;24(6):e00553-16. doi: 10.1128/CVI.00553-16. Print 2017 Jun. PMID 28446441
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 113866 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113866 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113866 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113866 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113866 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113866 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113866 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GSK2340272A Group | GSK2340269A Group
Started | 65 | 66
Completed | 64 | 65
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK2340272A Group | GSK2340269A Group | Total
Number analyzed (Participants) | 65 | 66 | 131
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.5 (14.29) | 38.4 (13.61) | 37.70 (13.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 35 | 78
  Male | 22 | 31 | 53
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Geographic ancestry: Asian-East Asian heritage | 0 | 1 | 1
  Geographic ancestry: White-Caucasian/European heritage | 65 | 65 | 130

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroconverted (SCR) Subjects for Hemagglutination Inhibition (HI) Antibodies Against Flu A/California/7/2009 (H1N1) Virus Strain
Description: Seroconversion was defined as: For initially seronegative subjects [antibody titer below (<) 10 post-vaccination], antibody titer greater than or equal to (≥) 40 after vaccination; For initially seropositive subjects (antibody titer ≥ 10 prior to vaccination), antibody titer after vaccination ≥ 4 fold the pre-vaccination antibody titer. The Flu strain assessed was A/California/7/2009 (H1N1)v-like influenza (Flu A/CAL/7/09).
Time Frame: At Day 21
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects who received 2 doses and for whom assay results were available for antibodies against H1N1 antigen for the blood sample taken 21 days after each vaccine dose.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 64 | 63
Participants | 60 | 44

2. Primary Outcome: Number of Subjects Who Were Seroprotected (SPR) for HI Antibodies Against the Flu A/California/7/2009 (H1N1) Virus Strain
Description: A seroprotected subject was defined as a vaccinated subject with a serum HI titer greater than or equal to (≥) 1:40, that usually is accepted as indicating protection.
Time Frame: At Day 21
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects who received 2 doses and for whom assay results were available for antibodies against H1N1 antigen for the blood sample taken 21 days after each vaccine dose.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 64 | 63
Participants | 60 | 46

3. Primary Outcome: Geometric Mean Fold Change (GMFR) for HI Antibodies Against Flu A/California/7/2009 (H1N1) Strain of Influenza Disease
Description: GMFR was defined as the fold change in serum HI geometric mean titers (GMTs) post-vaccination compared to pre-vaccination. The flu strain assessed was Flu A/CAL/7/09.
Time Frame: At Day 21
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 64 | 63
Fold change | 44.4 [33.6 to 58.7] | 11.4 [8.1 to 16.3]

4. Secondary Outcome: Number of Subjects Who Were Seropositive for Hemagglutination Inhibition (HI) Antibodies Against the Flu A/California/7/2009 (H1N1) Virus Strain
Description: A seropositive subject was defined as a vaccinated subject with a serum HI titer greater than or equal to (≥) 1:10, that usually is accepted as indicating protection.
Time Frame: At Days 0, 21 and 42
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 29 | 20
Participants
  Flu A/CAL/7/09, Day 0 | 29 | 20
  Flu A/CAL/7/09, Day 21 | 29 | 20
  Flu A/CAL/7/09, Day 42 | 29 | 20

5. Secondary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against the Flu A/California/7/2009 (H1N1) Strain of Influenza Disease
Description: Titers are presented as geometric mean titers (GMTs). The flu strain assessed was Flu A/CAL/7/09. The reference seropositivity cut-off value was ≥ 1:10.
Time Frame: At Days 0, 21 and 42
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 64 | 63
Titers
  Flu A/CAL/7/09, Day 0 | 9.6 [7.6 to 12.0] | 8.4 [6.7 to 10.6]
  Flu A/CAL/7/09, Day 21 | 424.0 [312.4 to 575.5] | 96.4 [64.0 to 145.3]
  Flu A/CAL/7/09, Day 42 | 686.7 [567.0 to 831.7] | 149.7 [108.0 to 207.7]

6. Secondary Outcome: Number of Subjects Who Were Seropositive for HI Antibodies Against Flu A/California/7/2009 (H1N1) Virus Strain
Description: A seropositive subject was defined as a vaccinated subject with a serum HI titer ≥ 1:10, that usually is accepted as indicating protection.
Time Frame: At Days 0, 21 and 42
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- GSK2340272A (18-40y): Healthy male or female adults, 18 to 40 years (18-40y) of age, who received two doses of GSK2340272A vaccine, administered intramuscularly in the deltoid region of the non-dominant arm at Day 0 and of the dominant arm at Day 21.
- GSK2340269A (18-40y): Healthy male or female adults, 18 to 40 years (18-40y) of age, who received two doses of GSK2340269A vaccine, administered intramuscularly in the deltoid region of the non-dominant arm at Day 0 and of the dominant arm at Day 21.
- GSK2340272A (41-60y): Healthy male or female adults, 41 to 60 years (41-60y) of age, who received two doses of GSK2340272A vaccine, administered intramuscularly in the deltoid region of the non-dominant arm at Day 0 and of the dominant arm at Day 21.
- GSK2340269A (41-60y): Healthy male or female adults, 41 to 60 years (41-60y) of age, who received two doses of GSK2340269A vaccine, administered intramuscularly in the deltoid region of the non-dominant arm at Day 0 and of the dominant arm at Day 21.
- GSK2340272A (41-50y): Healthy male or female adults, 41 to 50 years (41-50y) of age, who received two doses of GSK2340272A vaccine, administered intramuscularly in the deltoid region of the non-dominant arm at Day 0 and of the dominant arm at Day 21.
- GSK2340269A (41-50y): Healthy male or female adults, 41 to 50 years (41-50y) of age, who received two doses of GSK2340269A vaccine, administered intramuscularly in the deltoid region of the non-dominant arm at Day 0 and of the dominant arm at Day 21.
- GSK2340272A (51-60y): Healthy male or female adults, 51 to 60 years (15-60y) of age, who received two doses of GSK2340272A vaccine, administered intramuscularly in the deltoid region of the non-dominant arm at Day 0 and of the dominant arm at Day 21.
- GSK2340269A (51-60y): Healthy male or female adults, 41 to 60 years (51-60y) of age, who received two doses of GSK2340269A vaccine, administered intramuscularly in the deltoid region of the non-dominant arm at Day 0 and of the dominant arm at Day 21.
Arm/Group | GSK2340272A (18-40y) | GSK2340269A (18-40y) | GSK2340272A (41-60y) | GSK2340269A (41-60y) | GSK2340272A (41-50y) | GSK2340269A (41-50y) | GSK2340272A (51-60y) | GSK2340269A (51-60y)
Number analyzed (Participants) | 17 | 13 | 12 | 7 | 4 | 5 | 8 | 2
Participants
  Flu A/CAL/7/09, Day 0 | 17 | 13 | 12 | 7 | 4 | 5 | 8 | 2
  Flu A/CAL/7/09, Day 21 | 17 | 13 | 12 | 7 | 4 | 5 | 8 | 2
  Flu A/CAL/7/09, Day 42 | 17 | 13 | 12 | 7 | 4 | 5 | 8 | 2

7. Secondary Outcome: Titers for Serum HI Antibodies Against Flu A/California/7/2009 (H1N1) Strain of Influenza Disease
Description: as for outcome 5
Time Frame: At Days 0, 21 and 42
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2340272A (18-40y) | GSK2340269A (18-40y) | GSK2340272A (41-60y) | GSK2340269A (41-60y) | GSK2340272A (41-50y) | GSK2340269A (41-50y) | GSK2340272A (51-60y) | GSK2340269A (51-60y)
Number analyzed (Participants) | 32 | 31 | 32 | 32 | 16 | 16 | 16 | 16
Titers
  Flu A/CAL/7/09, Day 0 | 12.4 [8.2 to 18.7] | 10.9 [7.2 to 16.5] | 7.4 [6.1 to 8.9] | 6.5 [5.3 to 8.1] | 6.3 [5.0 to 8.1] | 7.5 [5.1 to 11.2] | 8.6 [6.3 to 11.7] | 5.7 [4.7 to 6.9]
  Flu A/CAL/7/09, Day 21 | 705.7 [523.8 to 950.7] | 171.1 [96.7 to 302.8] | 254.8 [156.7 to 414.4] | 55.4 [32.0 to 95.7] | 287.1 [164.1 to 502.1] | 123.3 [59.5 to 255.5] | 226.2 [95.3 to 536.6] | 24.8 [12.9 to 47.9]
  Flu A/CAL/7/09, Day 42 | 895.4 [714.7 to 1121.8] | 216.2 [134.8 to 346.8] | 526.7 [393.1 to 705.6] | 104.9 [67.4 to 163.2] | 462.5 [340.9 to 627.5] | 170.8 [94.4 to 308.8] | 599.7 [352.3 to 1020.8] | 64.4 [34.6 to 120.0]

8. Secondary Outcome: Number of Subjects Who Were Seropositive for HI Antibodies Against the Flu A/California/7/2009 (H1N1) Virus Strain
Description: as for outcome 4
Time Frame: At Days 182 and 364
Population: The analysis was performed on the ATP cohort for persistence at Day 182 and 364, which included all evaluable subjects who had received at least one dose of study vaccine according to their assignment, for whom data concerning immunogenicity outcome measures were available.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 64 | 63
Participants
  Flu A/CAL/7/09, Day 182 | 64 | 59
  Flu A/CAL/7/09, Day 364: number analyzed (Participants) | 61 | 61
  Flu A/CAL/7/09, Day 364 | 60 | 49

9. Secondary Outcome: Titers for Serum HI Antibodies Against the Flu A/California/7/2009 (H1N1) Strain of Influenza Disease
Description: Titers are presented as geometric mean titers (GMTs). The flu strain assessed was Flu A/CAL/7/09. The reference seropositivity cut-off value was greater than or equal to (≥) 1:10.
Time Frame: At Days 182 and 364
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 64 | 63
Titers
  Flu A/CAL/7/09, Day 182 | 222.6 [172.4 to 287.4] | 80.4 [55.1 to 117.2]
  Flu A/CAL/7/09, Day 364: number analyzed (Participants) | 61 | 61
  Flu A/CAL/7/09, Day 364 | 76.8 [58.1 to 101.5] | 35.2 [24.0 to 51.7]

10. Secondary Outcome: Number of Subjects Who Were Seropositive for HI Antibodies Against Flu A/California/7/2009 (H1N1) Virus Strain
Description: as for outcome 6
Time Frame: At Days 182 and 364
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A (18-40y) | GSK2340269A (18-40y) | GSK2340272A (41-50y) | GSK2340269A (41-50y) | GSK2340272A (51-60y) | GSK2340269A (51-60y)
Number analyzed (Participants) | 32 | 31 | 16 | 16 | 16 | 16
Participants
  Flu A/CAL/7/09, Day 182 | 32 | 29 | 16 | 16 | 16 | 14
  Flu A/CAL/7/09, Day 364: number analyzed (Participants) | 30 | 29 | 16 | 16 | 15 | 16
  Flu A/CAL/7/09, Day 364 | 30 | 26 | 16 | 14 | 14 | 9

11. Secondary Outcome: Titers for Serum HI Antibodies Against Flu A/California/7/2009 (H1N1) Strain of Influenza Disease
Description: as for outcome 5
Time Frame: At Days 182 and 364
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2340272A (18-40y) | GSK2340269A (18-40y) | GSK2340272A (41-50y) | GSK2340269A (41-50y) | GSK2340272A (51-60y) | GSK2340269A (51-60y)
Number analyzed (Participants) | 32 | 31 | 16 | 16 | 16 | 16
Titers
  Flu A/CAL/7/09, Day 182 | 269.1 [183.9 to 393.9] | 132.3 [75.9 to 230.4] | 182.2 [126.8 to 261.7] | 99.3 [47.8 to 206.6] | 186.1 [97.5 to 355.4] | 24.8 [15.6 to 39.6]
  Flu A/CAL/7/09, Day 364: number analyzed (Participants) | 30 | 29 | 16 | 16 | 15 | 16
  Flu A/CAL/7/09, Day 364 | 96.2 [63.1 to 146.7] | 57.2 [32.2 to 101.8] | 57.7 [38.4 to 86.8] | 48.4 [23.2 to 101.1] | 66.4 [33.1 to 133.2] | 10.6 [6.8 to 16.7]

12. Secondary Outcome: Number of Seroconverted (SCR) Subjects for HI Antibodies Against Flu A/California/7/2009 (H1N1) Strain of Influenza Disease
Description: as for outcome 1
Time Frame: At Days 21 and 42
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A (18-40y) | GSK2340269A (18-40y) | GSK2340272A (41-50y) | GSK2340269A (41-50y) | GSK2340272A (51-60y) | GSK2340269A (51-60y)
Number analyzed (Participants) | 32 | 31 | 16 | 16 | 16 | 16
Participants
  Flu A/CAL/7/09, Day 21 | 32 | 25 | 16 | 12 | 12 | 7
  Flu A/CAL/7/09, Day 42 | 32 | 27 | 16 | 15 | 16 | 12

13. Secondary Outcome: Number of Seroconverted (SCR) Subjects for HI Antibodies Against the Flu A/California/7/2009 (H1N1) Strain of Influenza Disease
Description: as for outcome 1
Time Frame: At Days 182 and 364
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 64 | 63
Participants
  Flu A/CAL/7/09, Day 182 | 60 | 42
  Flu A/CAL/7/09, Day 364: number analyzed (Participants) | 61 | 61
  Flu A/CAL/7/09, Day 364 | 44 | 22

14. Secondary Outcome: Number of Seroconverted (SCR) Subjects for HI Antibodies Against Flu A/California/7/2009 (H1N1) Strain of Influenza Disease
Description: Seroconversion was defined as: For initially seronegative subjects (antibody titer < 10 post-vaccination), antibody titer ≥ 40 after vaccination; For initially seropositive subjects (antibody titer ≥ 10 prior to vaccination), antibody titer after vaccination ≥ 4 fold the pre-vaccination antibody titer. The Flu strain assessed was A/California/7/2009 (H1N1)v-like influenza (Flu A/CAL/7/09).
Time Frame: At Days 182 and 364
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A (18-40y) | GSK2340269A (18-40y) | GSK2340272A (41-50y) | GSK2340269A (41-50y) | GSK2340272A (51-60y) | GSK2340269A (51-60y)
Number analyzed (Participants) | 32 | 31 | 16 | 16 | 16 | 16
Participants
  Flu A/CAL/7/09, Day 182 | 30 | 25 | 16 | 11 | 14 | 6
  Flu A/CAL/7/09, Day 364: number analyzed (Participants) | 30 | 29 | 16 | 16 | 15 | 16
  Flu A/CAL/7/09, Day 364 | 23 | 14 | 11 | 6 | 10 | 2

15. Secondary Outcome: Number of Subjects Who Were Seroprotected (SPR) for HI Antibodies Against the Flu A/California/7/2009 (H1N1) Virus Strain
Description: as for outcome 2
Time Frame: At Days 0, 21 and 42
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A (18-40y) | GSK2340269A (18-40y) | GSK2340272A (41-60y) | GSK2340269A (41-60y) | GSK2340272A (41-50y) | GSK2340269A (41-50y) | GSK2340272A (51-60y) | GSK2340269A (51-60y)
Number analyzed (Participants) | 32 | 31 | 32 | 32 | 16 | 16 | 16 | 16
Participants
  Flu A/CAL/7/09, Day 0 | 7 | 5 | 0 | 1 | 0 | 1 | 0 | 0
  Flu A/CAL/7/09, Day 21 | 32 | 26 | 28 | 20 | 16 | 13 | 12 | 7
  Flu A/CAL/7/09, Day 42 | 32 | 28 | 32 | 28 | 16 | 16 | 16 | 12

16. Secondary Outcome: Number of Subjects Who Were Seroprotected (SPR) for HI Antibodies Against the Flu A/California/7/2009 (H1N1) Virus Strain
Description: A seroprotected subject was defined as a vaccinated subject with a serum HI titer ≥ 1:40, that usually is accepted as indicating protection.
Time Frame: At Days 182 and 364
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A (18-40y) | GSK2340269A (18-40y) | GSK2340272A (41-50y) | GSK2340269A (41-50y) | GSK2340272A (51-60y) | GSK2340269A (51-60y)
Number analyzed (Participants) | 32 | 31 | 16 | 16 | 16 | 16
Participants
  Flu A/CAL/7/09, Day 182 | 32 | 26 | 16 | 12 | 14 | 7
  Flu A/CAL/7/09, Day 364: number analyzed (Participants) | 30 | 29 | 16 | 16 | 15 | 16
  Flu A/CAL/7/09, Day 364 | 26 | 17 | 11 | 7 | 11 | 2

17. Secondary Outcome: Geometric Mean Fold Change (GMFR) for HI Antibodies Against Flu A/California/7/2009 (H1N1) Strain of Influenza Disease
Description: as for outcome 3
Time Frame: At Days 21 and 42
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | GSK2340272A (18-40y) | GSK2340269A (18-40y) | GSK2340272A (41-50y) | GSK2340269A (41-50y) | GSK2340272A (51-60y) | GSK2340269A (51-60y)
Number analyzed (Participants) | 32 | 31 | 16 | 16 | 16 | 16
Fold change
  Flu A/CAL/7/09, Day 21 | 56.9 [38.9 to 83.4] | 15.7 [9.6 to 25.6] | 45.3 [27.8 to 73.6] | 16.4 [7.9 to 33.9] | 26.4 [13.2 to 52.9] | 4.4 [2.4 to 8.0]
  Flu A/CAL/7/09, Day 42 | 72.2 [49.3 to 105.9] | 19.8 [13.2 to 29.7] | 72.9 [52.9 to 100.6] | 22.7 [11.9 to 43.1] | 70.1 [41.9 to 117.4] | 11.3 [6.1 to 20.9]

18. Secondary Outcome: Geometric Mean Fold Change (GMFR) for HI Antibodies Against Flu A/California/7/2009 (H1N1) Strain of Influenza Disease
Description: as for outcome 3
Time Frame: At Days 182 and 364
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | GSK2340272A (18-40y) | GSK2340269A (18-40y) | GSK2340272A (41-50y) | GSK2340269A (41-50y) | GSK2340272A (51-60y) | GSK2340269A (51-60y)
Number analyzed (Participants) | 32 | 31 | 16 | 16 | 16 | 16
Fold change
  Flu A/CAL/7/09, Day 182 | 21.7 [15.4 to 30.6] | 12.1 [7.7 to 19.0] | 28.7 [19.1 to 43.2] | 13.2 [6.3 to 27.6] | 21.8 [12.7 to 37.2] | 4.4 [2.8 to 6.8]
  Flu A/CAL/7/09, Day 364: number analyzed (Participants) | 30 | 29 | 16 | 16 | 15 | 16
  Flu A/CAL/7/09, Day 364 | 8.4 [5.5 to 12.8] | 5.6 [3.5 to 8.9] | 9.1 [5.7 to 14.5] | 6.4 [3.1 to 13.4] | 8.0 [4.7 to 13.8] | 1.9 [1.2 to 2.9]

19. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = significant pain at rest; prevented normal activities as assessed by inability to attend/do work or school. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site.
Time Frame: During the 7-day post-vaccination period following Dose 1 (Day 0-6), Dose 2 (Day 21-27), and across doses (Day 0-6 and 21-27)
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects who filled in their symptom sheets.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 65 | 66
Participants
  Any Pain, Dose 1 | 60 | 16
  Grade 3 Pain, Dose 1 | 1 | 0
  Any Redness, Dose 1 | 4 | 0
  Grade 3 Redness, Dose 1 | 0 | 0
  Any Swelling, Dose 1 | 8 | 0
  Grade 3 Swelling, Dose 1 | 0 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 64 | 64
  Any Pain, Dose 2 | 57 | 11
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 64 | 64
  Grade 3 Pain, Dose 2 | 1 | 0
  Any Redness, Dose 2: number analyzed (Participants) | 64 | 64
  Any Redness, Dose 2 | 6 | 0
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 64 | 64
  Grade 3 Redness, Dose 2 | 0 | 0
  Any Swelling, Dose 2: number analyzed (Participants) | 64 | 64
  Any Swelling, Dose 2 | 6 | 0
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 64 | 64
  Grade 3 Swelling, Dose 2 | 0 | 0
  Any Pain, Across doses | 62 | 21
  Grade 3 Pain, Across doses | 1 | 0
  Any Redness, Across doses | 9 | 0
  Grade 3 Redness, Across doses | 0 | 0
  Any Swelling, Across doses | 11 | 0
  Grade 3 Swelling, Across doses | 0 | 0

20. Secondary Outcome: Number of Days With Solicited Local Symptoms
Description: The number of days with any solicited local symptoms reported during the solicited post-vaccination period. No subjects in GSK2340269A Group reported redness or swelling.
Time Frame: as for outcome 19
Population: as for outcome 19
Measure: Median (Inter-Quartile Range); unit: Days
Units Other Than Participants: Doses with the symptom
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 65 | 66
Number analyzed (Doses with the symptom) | 117 | 27
Days
  Pain, Dose 1: number analyzed (Doses with the symptom) | 60 | 16
  Pain, Dose 1 | 3.0 [3.0 to 4.0] | 2.0 [1.0 to 2.0]
  Pain, Dose 2: number analyzed (Doses with the symptom) | 57 | 11
  Pain, Dose 2 | 3.0 [2.0 to 4.0] | 2.0 [1.0 to 2.0]
  Pain, Overall/dose | 3.0 [2.0 to 4.0] | 2.0 [1.0 to 2.0]
  Redness, Dose 1: number analyzed (Doses with the symptom) | 4 | 0
  Redness, Dose 1 | 2.0 [1.5 to 2.5] |
  Redness, Dose 2: number analyzed (Doses with the symptom) | 6 | 0
  Redness, Dose 2 | 2.5 [2.0 to 4.0] |
  Redness, Overall/dose: number analyzed (Doses with the symptom) | 10 | 0
  Redness, Overall/dose | 2.0 [2.0 to 3.0] |
  Swelling, Dose 1: number analyzed (Doses with the symptom) | 8 | 0
  Swelling, Dose 1 | 1.5 [1.0 to 2.5] |
  Swelling, Dose 2: number analyzed (Doses with the symptom) | 9 | 0
  Swelling, Dose 2 | 2.0 [2.0 to 3.0] |
  Swelling, Overall/dose: number analyzed (Doses with the symptom) | 14 | 0
  Swelling, Overall/dose | 2.0 [1.0 to 3.0] |

21. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, headache, joint pain at other location, muscle aches, shivering, sweating and fever [defined as axillary temperature equal to or above (≥) 37.5 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade or their relationship to vaccination. Grade 3 symptom = general symptom that prevented normal everyday activities as assessed by inability to attend/do work or school, or required intervention of a physician/healthcare provider. Grade 3 fever = temperature ≥ 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: as for outcome 19
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 65 | 66
Participants
  Any Fatigue, Dose 1 | 31 | 22
  Grade 3 Fatigue, Dose 1 | 0 | 2
  Related Fatigue, Dose 1 | 28 | 18
  Any Headache, Dose 1 | 25 | 16
  Grade 3 Headache, Dose 1 | 1 | 0
  Related Headache, Dose 1 | 22 | 11
  Any Joint pain, Dose 1 | 13 | 4
  Grade 3 Joint pain, Dose 1 | 1 | 1
  Related Joint pain, Dose 1 | 12 | 2
  Any Muscle aches, Dose 1 | 17 | 6
  Grade 3 Muscle aches, Dose 1 | 1 | 1
  Related Muscle aches, Dose 1 | 16 | 5
  Any Shivering, Dose 1 | 9 | 6
  Grade 3 Shivering, Dose 1 | 0 | 1
  Related Shivering, Dose 1 | 9 | 6
  Any Sweating, Dose 1 | 9 | 9
  Grade 3 Sweating, Dose 1 | 0 | 1
  Related Sweating, Dose 1 | 8 | 9
  Any Temperature, Dose 1 | 2 | 2
  Grade 3 Temperature, Dose 1 | 0 | 0
  Related Temperature, Dose 1 | 1 | 2
  Any Fatigue, Dose 2: number analyzed (Participants) | 64 | 64
  Any Fatigue, Dose 2 | 28 | 15
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 64 | 64
  Grade 3 Fatigue, Dose 2 | 2 | 0
  Related Fatigue, Dose 2: number analyzed (Participants) | 64 | 64
  Related Fatigue, Dose 2 | 27 | 13
  Any Headache, Dose 2: number analyzed (Participants) | 64 | 64
  Any Headache, Dose 2 | 21 | 10
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 64 | 64
  Grade 3 Headache, Dose 2 | 0 | 0
  Related Headache, Dose 2: number analyzed (Participants) | 64 | 64
  Related Headache, Dose 2 | 20 | 9
  Any Joint pain, Dose 2: number analyzed (Participants) | 64 | 64
  Any Joint pain, Dose 2 | 12 | 1
  Grade 3 Joint pain, Dose 2: number analyzed (Participants) | 64 | 64
  Grade 3 Joint pain, Dose 2 | 0 | 0
  Related Joint pain, Dose 2: number analyzed (Participants) | 64 | 64
  Related Joint pain, Dose 2 | 12 | 1
  Any Muscle aches, Dose 2: number analyzed (Participants) | 64 | 64
  Any Muscle aches, Dose 2 | 22 | 3
  Grade 3 Muscle aches, Dose 2: number analyzed (Participants) | 64 | 64
  Grade 3 Muscle aches, Dose 2 | 0 | 0
  Related Muscle aches, Dose 2: number analyzed (Participants) | 64 | 64
  Related Muscle aches, Dose 2 | 22 | 1
  Any Shivering, Dose 2: number analyzed (Participants) | 64 | 64
  Any Shivering, Dose 2 | 12 | 2
  Grade 3 Shivering, Dose 2: number analyzed (Participants) | 64 | 64
  Grade 3 Shivering, Dose 2 | 0 | 0
  Related Shivering, Dose 2: number analyzed (Participants) | 64 | 64
  Related Shivering, Dose 2 | 12 | 2
  Any Sweating, Dose 2: number analyzed (Participants) | 64 | 64
  Any Sweating, Dose 2 | 8 | 4
  Grade 3 Sweating, Dose 2: number analyzed (Participants) | 64 | 64
  Grade 3 Sweating, Dose 2 | 0 | 0
  Related Sweating, Dose 2: number analyzed (Participants) | 64 | 64
  Related Sweating, Dose 2 | 8 | 4
  Any Temperature, Dose 2: number analyzed (Participants) | 64 | 64
  Any Temperature, Dose 2 | 1 | 0
  Grade 3 Temperature, Dose 2: number analyzed (Participants) | 64 | 64
  Grade 3 Temperature, Dose 2 | 0 | 0
  Related Temperature, Dose 2: number analyzed (Participants) | 64 | 64
  Related Temperature, Dose 2 | 1 | 0
  Any Fatigue, Across doses | 38 | 30
  Grade 3 Fatigue, Across doses | 2 | 2
  Related Fatigue, Across doses | 35 | 27
  Any Headache, Across doses | 37 | 22
  Grade 3 Headache, Across doses | 1 | 0
  Related Headache, Across doses | 35 | 18
  Any Joint pain, Across doses | 22 | 5
  Grade 3 Joint pain, Across doses | 1 | 1
  Related Joint pain, Across doses | 21 | 3
  Any Muscle aches, Across doses | 32 | 9
  Grade 3 Muscle aches, Across doses | 1 | 1
  Related Muscle aches, Across doses | 31 | 6
  Any Shivering, Across doses | 17 | 7
  Grade 3 Shivering, Across doses | 0 | 1
  Related Shivering, Across doses | 17 | 7
  Any Sweating, Across doses | 15 | 12
  Grade 3 Sweating, Across doses | 0 | 1
  Related Sweating, Across doses | 15 | 12
  Any Temperature, Across doses | 3 | 2
  Grade 3 Temperature, Across doses | 0 | 0
  Related Temperature, Across doses | 2 | 2

22. Secondary Outcome: Number of Days With Solicited General Symptoms
Description: The number of days with any solicited general symptoms reported during the solicited post-vaccination period. No subjects from the GSK2340269A Group reported any temperature after Dose 2.
Time Frame: as for outcome 19
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Median (Inter-Quartile Range); unit: Days
Units Other Than Participants: Doses with the symptom
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 65 | 66
Number analyzed (Doses with the symptom) | 59 | 37
Days
  Fatigue, Dose 1: number analyzed (Doses with the symptom) | 31 | 22
  Fatigue, Dose 1 | 2.0 [1.0 to 3.0] | 2.0 [2.0 to 4.0]
  Fatigue, Dose 2: number analyzed (Doses with the symptom) | 28 | 15
  Fatigue, Dose 2 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 4.0]
  Fatigue, Overall/dose | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 4.0]
  Headache, Dose 1: number analyzed (Doses with the symptom) | 25 | 16
  Headache, Dose 1 | 2.0 [1.0 to 3.0] | 1.5 [1.0 to 2.0]
  Headache, Dose 2: number analyzed (Doses with the symptom) | 21 | 10
  Headache, Dose 2 | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 2.0]
  Headache, Overall/dose: number analyzed (Doses with the symptom) | 46 | 26
  Headache, Overall/dose | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 2.0]
  Joint pain, Dose 1: number analyzed (Doses with the symptom) | 13 | 4
  Joint pain, Dose 1 | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0]
  Joint pain, Dose 2: number analyzed (Doses with the symptom) | 12 | 1
  Joint pain, Dose 2 | 2.0 [1.0 to 2.0] | 2.0 [2.0 to 2.0]
  Joint pain, Overall/dose: number analyzed (Doses with the symptom) | 25 | 5
  Joint pain, Overall/dose | 2.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0]
  Muscle aches, Dose 1: number analyzed (Doses with the symptom) | 17 | 6
  Muscle aches, Dose 1 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Muscle aches, Dose 2: number analyzed (Doses with the symptom) | 22 | 3
  Muscle aches, Dose 2 | 2.0 [1.0 to 3.0] | 1.0 [1.0 to 2.0]
  Muscle aches, Overall/dose: number analyzed (Doses with the symptom) | 39 | 9
  Muscle aches, Overall/dose | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 2.0]
  Sweating, Dose 1: number analyzed (Doses with the symptom) | 9 | 9
  Sweating, Dose 1 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Sweating, Dose 2: number analyzed (Doses with the symptom) | 8 | 4
  Sweating, Dose 2 | 2.0 [1.0 to 4.0] | 2.0 [2.0 to 2.5]
  Sweating, Overall/dose: number analyzed (Doses with the symptom) | 17 | 13
  Sweating, Overall/dose | 2.0 [1.0 to 4.0] | 2.0 [1.0 to 3.0]
  Shivering, Dose 1: number analyzed (Doses with the symptom) | 9 | 6
  Shivering, Dose 1 | 1.0 [1.0 to 2.0] | 1.5 [1.0 to 4.0]
  Shivering, Dose 2: number analyzed (Doses with the symptom) | 12 | 2
  Shivering, Dose 2 | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 3.0]
  Shivering, Overall/dose: number analyzed (Doses with the symptom) | 21 | 8
  Shivering, Overall/dose | 1.0 [1.0 to 2.0] | 1.5 [1.0 to 3.5]
  Temperature, Dose 1: number analyzed (Doses with the symptom) | 2 | 2
  Temperature, Dose 1 | 1.5 [1.0 to 2.0] | 1.5 [1.0 to 2.0]
  Temperature, Dose 2: number analyzed (Doses with the symptom) | 1 | 0
  Temperature, Dose 2 | 1.0 [1.0 to 1.0] |
  Temperature, Overall/dose: number analyzed (Doses with the symptom) | 3 | 2
  Temperature, Overall/dose | 1.0 [1.0 to 2.0] | 1.5 [1.0 to 2.0]

23. Secondary Outcome: Number of Subjects With Adverse Events of Specific Interest (AESIs)
Description: An AESI was defined as an AE including autoimmune diseases and other mediated inflammatory disorders and assessed by the investigator as specific to the treatment administration.
Time Frame: From Day 0 up to Day 364
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Groups:
- GSK2340269A Group: New Group 2 Description
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 65 | 66
Participants | 0 | 0

24. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: Within 21 days after the first vaccination and 63 days after the second vaccination (Day 0 - Day 20 and Day 21 - Day 84)
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 65 | 66
Participants
  Any AE(s), Days 0-20 | 25 | 25
  Grade 3 AE(s), Days 0-20 | 1 | 3
  Related AE(s), Days 0-20 | 11 | 7
  Any AE(s), up to Day 84 | 48 | 39
  Grade 3 AE(s), up to Day 84 | 7 | 9
  Related AE(s), up to Day 84 | 15 | 10

25. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study period (from Day 0 up to Day 364)
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 65 | 66
Participants | 4 | 4

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 7-day (Days 0-6) post-vaccination period; Unsolicited AEs: within the 84-day (Days 0-83) post-vaccination period; SAEs: during the entire study period (from Day 0 up to Day 364).
Arm/Group | GSK2340272A Group | GSK2340269A Group
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/66
Serious Adverse Events (participants affected / at risk) | 4/65 | 4/66
Other Adverse Events (participants affected / at risk) | 63/65 | 51/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK2340272A Group (N=65) | GSK2340269A Group (N=66)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Abortion spontaneous complete (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Balance disorder (Nervous system disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal disorder (Renal and urinary disorders) | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1
Open wound (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK2340272A Group (N=65) | GSK2340269A Group (N=66)
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 (27) | 7 (8)
Chills (General disorders) | 17 (21) | 7 (8)
Erythema (Skin and subcutaneous tissue disorders) | 9 (10) | 0 (0)
Fatigue (General disorders) | 38 (60) | 31 (41)
Gastroenteritis (Infections and infestations) | 4 (4) | 3 (3)
Headache (Nervous system disorders) | 39 (53) | 24 (30)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 15 (17) | 12 (13)
Influenza like illness (General disorders) | 3 (3) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 32 (40) | 9 (9)
Pain (General disorders) | 62 (117) | 21 (27)
Pyrexia (General disorders) | 5 (5) | 4 (4)
Rhinitis (Infections and infestations) | 3 (3) | 6 (6)
Swelling (General disorders) | 11 (14) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 14 (14) | 8 (8)
Redness (General disorders) | 9 | 0
Joint Pain ar other location (General disorders) | 22 | 5
Muscle aches (General disorders) | 32 | 9
Shivering (General disorders) | 17 | 7
Sweating (General disorders) | 15 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.